CLINICAL TRIAL: NCT04169503
Title: Immune Checkpoint Inhibitors Rechallenge After Immune-related Adverse Events in Patients With Cancer: an Observational and Retrospective Study Using the WHO Pharmacovigilance Database
Brief Title: Immune Checkpoint Inhibitors Rechallenge After Immune-related Adverse Events
Acronym: 19-916
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco15-19-07
Record Dates: First submitted 2019-07-19; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Immune Checkpoint Modulator — identification of cases of immune-related adverse events due to immune checkpoint inhibitors. Among these cases, identification and description of those with immune checkpoint inhibitor rechallenge.

SUMMARY:
Although immune checkpoint inhibitors (ICIs) have proved effective in treating many cancers, patients receiving ICIs may experience immune-related adverse events (irAEs). Little evidence exists on the safety of resuming these treatments after an irAE.

Our objective was to investigate the safety of ICI rechallenge after an irAE using the WHO pharmacovigilance database

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database (VigiBase) of individual safety case reports at the time of the extraction,
* consecutive individual case safety reports present in VigiBase reporting an irAEs associated to at least one immune checkpoint inhibitor.

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with immune checkpoint inhibitors and experiencing irAEs
Sampling Method: Non-Probability Sample
Enrollment: 17562 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of second immune-related adverse events (irAEs) | Number of case reported in the World Health Organization (WHO) of individual safety case reports, through study completion (an average of 2 months).
  percentage of cases experiencing a second irAE among the rechallenged cases

SECONDARY OUTCOMES:
Description of cases experiencing an initial irAEs | Number of case reported in the World Health Organization (WHO) of individual safety case reports, through study completion (an average of 2 months)..
  description of clinical features of cases experiencing an initial irAEs
Description of the rechallenge cases | Number of case reported in the World Health Organization (WHO) of individual safety case reports, through study completion (an average of 2 months)..
  description of clinical features of the rechallenged cases
Description of the clinical features of cases experiencing a second irAEs | Number of case reported in the World Health Organization (WHO) of individual safety case reports, through study completion (an average of 2 months)..
  Description of the clinical features of cases experiencing a second irAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France